CLINICAL TRIAL: NCT00002663
Title: An Evaluation of the Toxicity and Therapeutic Effects of Epstein-Barr Virus-Immune T-Lymphocytes Derived From a Normal HLA-Compatible or Haplotype-Matched Donor in the Treatment of EBV-Associated Lymphoproliferative Diseases or Malignancies and Patients With Detectable Circulating Levels of EBV DNA Who Are at High Risk for EBV-Associated Lymphoproliferative Diseases
Brief Title: Biological Therapy in Treating Patients at High-Risk or With Lymphoma, Lymphoproliferative Disease, or Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Atara Biotherapeutics (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 95-024; P30CA008748 (NIH); MSKCC-95024; NCI-V95-0685
Expanded Access: NCT02822495 (No longer available)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-01

CONDITIONS: EBV-induced Lymphomas; EBV-associated Malignancies; Transplant Patients With EBV Viremia at High Risk of Developing a Recurrent EBV Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; childhood Burkitt lymphoma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; stage II childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; T-cell large granular lymphocyte leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; AIDS-related peripheral/systemic lymphoma; HIV-associated Hodgkin lymphoma; stage I childhood small noncleaved cell lymphoma; stage I childhood large cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage II childhood large cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; contiguous stage II small lymphocytic lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Large Granular Lymphocytic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell

ARMS (10):
- EBV+ PTLD-HCT R/R Rituximab (Tab-cel Only) (Experimental): Patients with Epstein-Barr virus positive (EBV+) posttransplant lymphoproliferative disorders (PTLD) following hematopoietic cell transplant (HCT) who were relapse/refractory (R/R) to rituximab will receive IV infusion of tabelecleucel (tab-cel) at 1-5 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Epstein-Barr virus-specific cytotoxic T lymphocytes (EBV-CTLs)
- EBV+ PTLD-SOT R/R Rituximab + Chemo (Tab-cel Only) (Experimental): Patients with EBV+ PTLD following solid organ transplant (SOT) who were R/R to rituximab and chemotherapy will receive IV infusion of tabelecleucel at 1-5 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Epstein-Barr virus-specific cytotoxic T lymphocytes (EBV-CTLs)
- EBV+ AID-LPD (Tab-cel Only) (Experimental): Patients with EBV+ acquired immunodeficiency (AID) lymphoproliferative disorder (LPD) will receive IV infusion of tabelecleucel at 1-5 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Epstein-Barr virus-specific cytotoxic T lymphocytes (EBV-CTLs)
- EBV+ LMS (Tab-cel Only) (Experimental): Patients with EBV+ leiomyosarcoma (LMS) will receive IV infusion of tabelecleucel at 1-5 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Epstein-Barr virus-specific cytotoxic T lymphocytes (EBV-CTLs)
- EBV+ NPC (Tab-cel Only) (Experimental): Patients with EBV+ nasopharyngeal carcinoma (NPC) will receive IV infusion of tabelecleucel at 1-5 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Epstein-Barr virus-specific cytotoxic T lymphocytes (EBV-CTLs)
- EBV+ PTLD-HCT R/R Rituximab (EBV-CTLs Only) (Experimental): Patients with EBV+ following PTLD HCT who were R/R to rituximab or rituximab naive will receive IV infusion of transplant donor-derived EBV-cytotoxic T lymphocytes (CTLs) at 1-5 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Epstein-Barr virus-specific cytotoxic T lymphocytes (EBV-CTLs)
- EBV+ PTLD-SOT R/R Rituximab + Chemo (EBV-CTLs Only) (Experimental): Patients with EBV+ PTLD following SOT who were R/R to rituximab and chemotherapy will receive IV infusion of transplant donor-derived EBV-CTLs at 1-5 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Epstein-Barr virus-specific cytotoxic T lymphocytes (EBV-CTLs)
- EBV+ Viremia (EBV-CTLs Only) (Experimental): Patients with EBV+ viremia will receive IV infusion of transplant donor-derived EBV-CTLs at 1-5 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Epstein-Barr virus-specific cytotoxic T lymphocytes (EBV-CTLs)
- EBV+ PID-LPD (Tab-cel or EBV-CTLs) (Experimental): Patients with EBV+ primary immunodeficiency (PID) LPD will receive IV infusion of tabelecleucel or transplant donor-derived EBV- CTLs at 1-5 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Epstein-Barr virus-specific cytotoxic T lymphocytes (EBV-CTLs)
- EBV+ Lymphoma (Tab-cel or EBV-CTLs) (Experimental): Patients with EBV+ lymphoma will receive IV infusion of tabelecleucel or transplant donor-derived EBV-CTLs at 1-5 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Epstein-Barr virus-specific cytotoxic T lymphocytes (EBV-CTLs)

INTERVENTIONS:
Biological: Epstein-Barr virus-specific cytotoxic T lymphocytes (EBV-CTLs) — EBV-CTLs are cytotoxic T lymphocytes that specifically kill cells presenting EBV protein antigens including EBV-transformed B lymphocytes responsible for EBV-associated lymphomas and lymphoproliferative disorders.
  Other Names: tabelecleucel (tab-cel®, ATA129), allogeneic EBV-CTLs; transplant donor-derived EBV-CTLs

SUMMARY:
The purpose of this phase I/II trial is to study the side effects and best dose of biological therapy to treat patients at high-risk or with Epstein-Barr virus-associated lymphoma or lymphoproliferative disease.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented EBV antigen positive lymphoproliferative disease, lymphoma, or other EBV-associated malignancy OR
* Severely immunocompromised patients who develop blood levels of EBV DNA exceeding 500 copies/ml DNA, and are therefore at high risk for developing an EBV LPD

It is expected that five types of patients afflicted with EBV-associated lymphomas or lymphoproliferative diseases will be referred and will consent to participate in this trial. These are:

1. Patients developing or at risk for EBV lymphomas or lymphoproliferative disorders following an allogeneic marrow transplant.
2. Patients developing or at risk for EBV lymphomas or lymphoproliferative disorders following an allogeneic organ transplant.
3. Patients with AIDS developing EBV lymphomas or lymphoproliferative diseases as a consequence of the profound acquired immunodeficiency induced by HIV.
4. Patients who develop EBV lymphomas or lymphoproliferative diseases as a consequence of profound immunodeficiencies associated with a congenital immune deficit or acquired as a sequela of anti-neoplastic or immunosuppressive therapy.
5. Patients who develop other EBV-associated malignancies without pre-existing immune deficiency, including: EBV+ Hodgkin's and Non- Hodgkin's disease, EBV+ nasopharyngeal carcinoma, EBV+ hemophagocytic lymphohistiocytosis, or EBV+ leiomyosarcoma.

Exclusion Criteria:

The following patients will be excluded from this study:

* Moribund patients who, by virtue of heart, kidney, liver, lung, or neurologic dysfunction not related to lymphoma, are unlikely to survive the 6-8 weeks required for in vitro generation and expansion of the EBV-specific T cells to be used for therapy and the subsequent 3 weeks required to achieve an initial assessment of the effects of infusions of EBV-specific T cells.
* Pregnancy does not constitute a contraindication to infusions of EBV-specific T cells.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 1995-03 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minoti Hiremath, MD, Study Director — Atara Biotherapeutics
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Prockop S, Doubrovina E, Suser S, Heller G, Barker J, Dahi P, Perales MA, Papadopoulos E, Sauter C, Castro-Malaspina H, Boulad F, Curran KJ, Giralt S, Gyurkocza B, Hsu KC, Jakubowski A, Hanash AM, Kernan NA, Kobos R, Koehne G, Landau H, Ponce D, Spitzer B, Young JW, Behr G, Dunphy M, Haque S, Teruya-Feldstein J, Arcila M, Moung C, Hsu S, Hasan A, O'Reilly RJ. Off-the-shelf EBV-specific T cell immunotherapy for rituximab-refractory EBV-associated lymphoma following transplantation. J Clin Invest. 2020 Feb 3;130(2):733-747. doi: 10.1172/JCI121127. PMID 31689242

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 58 participants were treated. However, 1 participant was analyzed in 2 different arms due to treatment. This participant was counted in only 1 arm for Participant Flow results and was counted in each arm for Outcome Measures.
Groups:
- EBV+ PTLD-HCT R/R Rituximab (Tab-cel Only): Participants with Epstein-Barr virus positive (EBV+) posttransplant lymphoproliferative disorders (PTLD) hematopoietic cell transplant (HCT) who were relapse/refractory (R/R) to rituximab received IV infusion of tabelecleucel (Tab-cel) on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ PTLD-SOT R/R Rituximab + Chemo (Tab-cel Only): Participants with EBV+PTLD solid organ transplant (SOT) who were R/R to rituximab and chemotherapy received IV infusion of tabelecleucel on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ AID-LPD (Tab-cel Only): Participants with EBV+ acquired immunodeficiency (AID) lymphoproliferative disorder (LPD) received IV infusion of tabelecleucel on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ LMS (Tab-cel Only): Participants with EBV+ leiomyosarcoma (LMS) received IV infusion of tabelecleucel on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ NPC (Tab-cel Only): Participants with EBV+ nasopharyngeal carcinoma (NPC) received IV infusion of tabelecleucel on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ PTLD-HCT R/R Rituximab (EBV-CTLs Only): Participants with EBV+PTLD HCT who were R/R to rituximab or rituximab naive received donor-derived EBV cytotoxic T lymphocyte (CTL) on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ PTLD-SOT R/R Rituximab + Chemo (EBV-CTLs Only): Participants with EBV+PTLD SOT received donor-derived EBV-CTLs on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ Viremia (EBV-CTLs Only): Participants with EBV+ viremia received donor-derived EBV-CTLs on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+PID-LPD (Tab-cel or EBV-CTLs Only): Participants with EBV+ primary immunodeficiency (PID) LPD received IV infusion of tabelecleucel or donor-derived EBV- CTLs on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ Lymphoma (Tab-cel or EBV-CTLs Only): Participants with EBV+ lymphoma received IV infusion of tabelecleucel or donor-derived EBV- CTLs on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | EBV+ PTLD-HCT R/R Rituximab (Tab-cel Only) | EBV+ PTLD-SOT R/R Rituximab + Chemo (Tab-cel Only) | EBV+ AID-LPD (Tab-cel Only) | EBV+ LMS (Tab-cel Only) | EBV+ NPC (Tab-cel Only) | EBV+ PTLD-HCT R/R Rituximab (EBV-CTLs Only) | EBV+ PTLD-SOT R/R Rituximab + Chemo (EBV-CTLs Only) | EBV+ Viremia (EBV-CTLs Only) | EBV+PID-LPD (Tab-cel or EBV-CTLs Only) | EBV+ Lymphoma (Tab-cel or EBV-CTLs Only)
Started | 11 | 4 | 2 | 5 | 1 | 23 | 2 | 6 | 2 | 2
Completed | 4 | 2 | 1 | 3 | 0 | 8 | 1 | 4 | 0 | 0
Not Completed | 7 | 2 | 1 | 2 | 1 | 15 | 1 | 2 | 2 | 2
Not completed — Death | 4 | 1 | 1 | 0 | 0 | 13 | 0 | 1 | 1 | 1
Not completed — Lost to Follow-up | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least one dose of study treatment (tabelecleucel or EBV-CTLs). Results from arms with <= 3 participants (as shown in the participant flow) are being excluded due to the low numbers of participants; these low numbers pose a risk for participant re-identification in these rare indications of this single center study.
Groups:
- EBV+ PTLD-HCT R/R Rituximab (Tab-cel Only): Participants with EBV+ PTLD HCT who were R/R to rituximab received IV infusion of tabelecleucel on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ PTLD-SOT R/R Rituximab + Chemo (Tab-cel Only): Participants with EBV+PTLD SOT who were R/R to rituximab and chemotherapy received IV infusion of tabelecleucel on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ LMS (Tab-cel Only): Participants with EBV+ LMS received IV infusion of tabelecleucel on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ PTLD-HCT R/R Rituximab (EBV-CTLs Only): Participants with EBV+PTLD HCT who were R/R to rituximab or rituximab naive received donor-derived EBV-CTL on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | EBV+ PTLD-HCT R/R Rituximab (Tab-cel Only) | EBV+ PTLD-SOT R/R Rituximab + Chemo (Tab-cel Only) | EBV+ LMS (Tab-cel Only) | EBV+ PTLD-HCT R/R Rituximab (EBV-CTLs Only) | EBV+ Viremia (EBV-CTLs Only) | Total
Number analyzed (Participants) | 11 | 4 | 5 | 23 | 7 | 50
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 7 | 3 | 4 | 8 | 3 | 25
  =>18 years | 4 | 1 | 1 | 15 | 4 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 2 | 7 | 2 | 19
  Male | 4 | 3 | 3 | 16 | 5 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2 | 1 | 5
  Not Hispanic or Latino | 1 | 1 | 0 | 4 | 1 | 7
  Unknown or Not Reported | 10 | 3 | 3 | 17 | 5 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 2 | 1 | 6
  White | 6 | 1 | 3 | 18 | 5 | 33
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 1 | 2 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The ORR is defined as percentage of participants with best overall response of complete remission/response (CR) or partial remission/response (PR) based on investigator's assessment. For participants with clinically and/or radiologically evident EBV LPD or malignancies, CR is complete resolution of all clinical and radiologic evidence of lymphoma, confirmed by biopsy of the affected tissues when indicated, lasting for at least 3 weeks following completion of a cycle of tabelecleucel; and PR is a 50 % or greater reduction in the size of all lymphomatous lesions as determined by computed tomography (CT) or magnetic resonance imaging (MRI) measurements of tumor volume, which was maintained for at least 3 weeks following completion of a cycle of tabelecleucel. For participants without clinically and/or radiologically evident tumors with increasing levels of EBV DNA, CR is clearance of EBV without subsequent development of EBV+ LPD; and PR is at least a 10-fold decrease in EBV DNA levels.
Time Frame: From Day 1 through 251.1 months after Day 1 dose
Population: Full analysis set included all participants who received at least one dose of study treatment (tabelecleucel or EBV-CTLs). Results from arms with <= 3 participants (as shown in the participant flow) are excluded due to the low numbers of participants; these low numbers pose a risk for participant re-identification in these rare indications of this single center study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- EBV+ PTLD-HCT R/R Rituximab (Tab-cel Only): Participants with EBV+ PTLD following HCT who were R/R to rituximab received IV infusion of tabelecleucel on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ PTLD-SOT R/R Rituximab + Chemo (Tab-cel Only): Participants with EBV+PTLD following SOT who were R/R to rituximab and chemotherapy received IV infusion of tabelecleucel on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ LMS (Tab-cel Only): Participants with EBV+ following LMS received IV infusion of tabelecleucel on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ PTLD-HCT R/R Rituximab (EBV-CTLs Only): Participants with EBV+PTLD following HCT who were R/R to rituximab or rituximab naive received donor-derived EBV-CTL on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ Viremia (EBV-CTLs Only): Participants with EBV+ following viremia received donor-derived EBV-CTLs on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
Arm/Group | EBV+ PTLD-HCT R/R Rituximab (Tab-cel Only) | EBV+ PTLD-SOT R/R Rituximab + Chemo (Tab-cel Only) | EBV+ LMS (Tab-cel Only) | EBV+ PTLD-HCT R/R Rituximab (EBV-CTLs Only) | EBV+ Viremia (EBV-CTLs Only)
Number analyzed (Participants) | 11 | 4 | 5 | 23 | 7
Percentage of participants | 63.6 [30.8 to 89.1] | 50.0 [6.8 to 93.2] | 0 [0 to 52.2] | 43.5 [23.2 to 65.5] | 57.1 [18.4 to 90.1]

2. Secondary Outcome: Overall Survival (OS)
Description: The OS is defined as the time from the first dose of tabelecleucel or EBV-CTLs to the date of death due to any cause. The OS was estimated using Kaplan-Meier method.
Time Frame: From Day 1 through 251.1 months after Day 1 dose
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- EBV+ PTLD-HCT R/R Rituximab (EBV-CTLs Only): Participants with EBV+PTLD following HCT who were R/R to rituximab or rituximab naive received donor-derived EBV-CTLs on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
Arm/Group | EBV+ PTLD-HCT R/R Rituximab (Tab-cel Only) | EBV+ PTLD-SOT R/R Rituximab + Chemo (Tab-cel Only) | EBV+ LMS (Tab-cel Only) | EBV+ PTLD-HCT R/R Rituximab (EBV-CTLs Only) | EBV+ Viremia (EBV-CTLs Only)
Number analyzed (Participants) | 11 | 4 | 5 | 23 | 7
Months | 14.8 [0.9 to NA] — Upper limit of confidence interval is not estimable due to insufficient events being observed at the time of the analysis. | 84.8 [1.1 to 115.0] | NA [60.6 to NA] — Median and upper limit of confidence interval are not estimable due to insufficient events being observed at the time of the analysis. | 18.6 [1.5 to NA] — Upper limit of confidence interval is not estimable due to insufficient events being observed at the time of the analysis. | NA [2.5 to NA] — Median and upper limit of confidence interval are not estimable due to insufficient events being observed at the time of the analysis.

3. Secondary Outcome: OS Rate at 12 Months
Description: Percentage of participants with OS at 12 months are reported. The OS is defined as the time from the first dose of tabelecleucel or EBV-CTLs to the date of death due to any cause. The OS was estimated using Kaplan-Meier method.
Time Frame: From Day 1 through 12 months after Day 1 dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EBV+ PTLD-HCT R/R Rituximab (Tab-cel Only) | EBV+ PTLD-SOT R/R Rituximab + Chemo (Tab-cel Only) | EBV+ LMS (Tab-cel Only) | EBV+ PTLD-HCT R/R Rituximab (EBV-CTLs Only) | EBV+ Viremia (EBV-CTLs Only)
Number analyzed (Participants) | 11 | 4 | 5 | 23 | 7
Percentage of participants | 54.5 [22.9 to 78.0] | 75.0 [12.8 to 96.1] | 100.0 [100 to 100] | 52.2 [30.5 to 70.0] | 85.7 [33.4 to 97.9]

4. Secondary Outcome: OS Follow-up Time
Description: The OS at follow-up time are reported. The OS is defined as the time from the first dose of tabelecleucel or EBV-CTLs to the date of death due to any cause. The OS was estimated using Kaplan-Meier method.
Time Frame: From Day 1 through 251.1 months after Day 1 dose
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | EBV+ PTLD-HCT R/R Rituximab (Tab-cel Only) | EBV+ PTLD-SOT R/R Rituximab + Chemo (Tab-cel Only) | EBV+ LMS (Tab-cel Only) | EBV+ PTLD-HCT R/R Rituximab (EBV-CTLs Only) | EBV+ Viremia (EBV-CTLs Only)
Number analyzed (Participants) | 11 | 4 | 5 | 23 | 7
Months | 14.82 [0.5 to 88.9] | 63.56 [1.1 to 115.0] | 77.40 [29.5 to 109.3] | 18.63 [0.2 to 251.1] | 62.98 [2.5 to 91.3]

5. Secondary Outcome: Time to Response (TTR)
Description: The TTR was defined as the time from the date of the first dose of tabelecleucel or EBV-CTLs to the date of a PR or CR, whichever occurred first. For participants with clinically and/or radiologically evident EBV LPD or malignancies, CR was defined as complete resolution of all clinical and radiologic evidence of lymphoma, confirmed by biopsy of the affected tissues when indicated, lasting for at least 3 weeks following completion of a cycle of tabelecleucel or EBV-CTLs; and a PR was defined as a 50 % or greater reduction in the size of all lymphomatous lesions as determined by CT or MRI scan measurements of tumor volume, which was maintained for at least 3 weeks following completion of a cycle of tabelecleucel or EBV-CTLs. For participants without clinically and/or radiologically evident tumors with increasing levels of EBV DNA, CR was defined as clearance of EBV without subsequent development of EBV+ LPD; and PR was defined as at least a 10-fold decrease in EBV DNA levels.
Time Frame: From Day 1 through 251.1 months after Day 1 dose
Population: Full analysis set included all participants who received at least one dose of study treatment (tabelecleucel or EBV-CTLs). Participants who achieved CR or PR were analyzed for this outcome measure. Results from arms with <= 3 participants (as shown in the participant flow) are excluded due to the low numbers of participants; these low numbers pose a risk for participant re-identification in these rare indications of this single center study.
Measure: Median (Full Range); unit: Months
Arm/Group | EBV+ PTLD-HCT R/R Rituximab (Tab-cel Only) | EBV+ PTLD-SOT R/R Rituximab + Chemo (Tab-cel Only) | EBV+ LMS (Tab-cel Only) | EBV+ PTLD-HCT R/R Rituximab (EBV-CTLs Only) | EBV+ Viremia (EBV-CTLs Only)
Number analyzed (Participants) | 7 | 2 | 0 | 10 | 4
Months | 1.18 [0.8 to 2.4] | 6.74 [3.1 to 10.4] |  | 1.45 [0.6 to 5.1] | 1.22 [1.1 to 1.4]

6. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: The CBR was the proportion of participants who have achieved a CR, PR or SD assessed at least 28 days after first dose date of study drug. For participants with clinically and/or radiologically evident EBV LPD or malignancies, CR as complete resolution of all clinical and radiologic evidence of lymphoma, confirmed by biopsy of affected tissues when indicated, lasting for at least 3 weeks following completion of a cycle of tabelecleucel or EBVCTLs; and a PR as a >= 50% reduction in size of all lymphomatous lesions as determined by CT or MRI scan measurements of tumor volume, maintained for at least 3 weeks following completion of a cycle of tabelecleucel or EBV-CTLs. For participants without clinically and/or radiologically evident tumors with increasing levels of EBV DNA, CR as clearance of EBV without subsequent development of EBV+ LPD; and PR as at least a 10-fold decrease in EBV DNA levels. The CBR was included specifically as clinically meaningful for solid tumor, namely LMS.
Time Frame: From Day 1 through 251.1 months after Day 1 dose
Population: Full analysis set included all participants who received at least one dose of study treatment (tabelecleucel or EBV-CTLs). Participants who achieved CR, PR or SD were analyzed for this outcome measure. Results from arms with <= 3 participants (as shown in the participant flow) are excluded due to the low numbers of participants; these low numbers pose a risk for participant re-identification in these rare indications of this single center study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EBV+ PTLD-HCT R/R Rituximab (Tab-cel Only) | EBV+ PTLD-SOT R/R Rituximab + Chemo (Tab-cel Only) | EBV+ LMS (Tab-cel Only) | EBV+ PTLD-HCT R/R Rituximab (EBV-CTLs Only) | EBV+ Viremia (EBV-CTLs Only)
Number analyzed (Participants) | 11 | 4 | 5 | 23 | 7
Percentage of participants | 63.6 [30.8 to 89.1] | 75.0 [19.4 to 99.4] | 80.0 [28.4 to 99.5] | 47.8 [26.8 to 69.4] | 71.4 [29.0 to 96.3]

ADVERSE EVENTS:
Time Frame: From Day 1 through 251.1 months after Day 1 dose
Description: Combined AE data for all enrolled participants are reported because few arms had <=3 participants which poses a risk of participant identification with rare indications in this study. Treatment-emergent SAEs includes events collected retrospectively and prospectively per protocol. Non-serious AEs were not collected, hence reported as '0'. In participant flow, 'Deaths' are reported as a reason for study discontinuation, whereas in 'All-Cause Mortality' deaths due to any cause are reported.
Groups:
- Overall Total: All eligible participants with EBV+ received IV infusion of tabelecleucel or donor-derived EBV-CTL on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
Arm/Group | Overall Total
All-Cause Mortality (participants affected / at risk) | 32/58
Serious Adverse Events (participants affected / at risk) | 40/58
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Total (N=58)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4)
Haemolysis (Blood and lymphatic system disorders) | 1 (2)
Left ventricular dysfunction (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Hypopituitarism (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Anal ulcer (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Device related thrombosis (General disorders) | 1 (1)
Disease progression (General disorders) | 3 (4)
Oedema (General disorders) | 2 (2)
Pyrexia (General disorders) | 13 (14)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 2 (2)
Renal transplant failure (Immune system disorders) | 1 (1)
Serum sickness (Immune system disorders) | 1 (1)
Device related infection (Infections and infestations) | 8 (9)
Ear infection bacterial (Infections and infestations) | 1 (1)
Ear infection staphylococcal (Infections and infestations) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 4 (5)
Neutropenic infection (Infections and infestations) | 3 (4)
Otitis media (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia fungal (Infections and infestations) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (3)
Intracranial pressure increased (Nervous system disorders) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Seizure (Nervous system disorders) | 3 (3)
Mental status changes (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Venoocclusive disease (Vascular disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
In this investigator-led study, scans were only collected as clinically indicated in lieu of a defined schedule; therefore, disease assessment endpoints (duration of response, durable response rate, progression-free survival, time to progression) may not be reliable, hence not reported. Study 95-024 was designed for patient treatment and conducted mostly as investigator-sponsored, single-center until Atara assumed responsibility, then relevant data was transferred from the investigator to Atara.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT00002663/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT00002663/SAP_001.pdf